CLINICAL TRIAL: NCT06059066
Title: Optimization of OnabotulinumtoxinA (BTX-A) Injection for the Treatment of Neurogenic Lower Urinary Tract Dysfunction
Acronym: BOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Collaborating for Advancement of Interdisciplinary Research in Benign Urology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00037721
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-03

CONDITIONS: Neurogenic Bladder; Lower Urinary Tract Symptoms; Overactive Bladder; Neuro: Neurogenic Bladder; Neurogenic Detrusor Overactivity
Keywords: neurogenic bladder; Lower urinary tract symptoms; Neurogenic detrusor overactivity; Onabotulinum toxinA
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Lower Urinary Tract Symptoms; Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Injection Sites (Active Comparator): Standard number of injections
  Interventions: Procedure: Standard number of injection sites
- Reduced Injection Sites (Experimental): Reduced number of injections
  Interventions: Procedure: Reduced number of injection sites

INTERVENTIONS:
Procedure: Standard number of injection sites — 200 units or 300 units BTX-A reconstituted in 20 mL normal saline, injected into the bladder detrusor in 20 separate injections of 1 mL including the trigone.
  Arms: Standard Injection Sites
Procedure: Reduced number of injection sites — 200 units or 300 units BTX-A reconstituted in 5 mL normal saline, injected into the bladder detrusor in 5 separate injections of 1 mL including the trigone.
  Arms: Reduced Injection Sites

SUMMARY:
The purpose of this study is to evaluate and standardize the way providers perform OnabotulinumtoxinA (BTX-A) injections into the bladder for the diagnosis of neurogenic lower urinary tract dysfunction (NLUTD)/overactive bladder (OAB). NLUTD/OAB is a syndrome that affects many people, and includes urinary frequency, urinary urgency, urgency incontinence, and nocturia. This syndrome can be challenging to treat and often requires procedural management - including BTX-A injections into the bladder.

DETAILED DESCRIPTION:
Neurological disorders such as Multiple Sclerosis (MS), Spinal Cord Injury (SCI), Parkinson's Disease (PD), Spina Bifida (SB), and stroke disrupt neural control of voiding and lead to the development of neurogenic lower urinary tract dysfunction (NLUTD), which develops when either the detrusor muscle fails to maintain effective contractions (voiding phase) or fails to relax appropriately with low pressures (storage phase), if the urethral sphincter (internal or external) fails to lower its tonicity and resistance, or if there is an asynchrony in events eventually leading to detrusor sphincter dyssynergia (DSD). Different patterns of NLUTD (including both storage and voiding) can arise depending on the level of injury or type of neurological disease. It can be characterized by urinary urgency, frequency and incontinence or urinary hesitancy and retention that leads to urinary tract infections (UTIs). Some patients develop neurogenic overactive bladder (NOAB).

Management of NOAB symptoms is complex. Treatment with BTX-A has been shown to decrease episodes of urinary incontinence and improve quality of life in this population. It has also been shown to ameliorate a multitude of devastating complications, such as upper tract deterioration, recurrent urinary tract infections, sepsis, and death. According to the current manufacturer's recommendation, a standard 200-unit vial of Botox® should be diluted in 30cc of 0.9% saline and injected across 30 different sites in the detrusor muscle (Figure 2). Despite these guidelines, there are wide variations in administration techniques, raising the question what is the best depth and location for injection, and optimal concentration and volume of toxin per injection site. The objective of this study is to determine the optimal injection schema for 200 units or more of intradetrusor BTX-A in patients with NOAB in the office setting.

The investigators hypothesize that patients with NOAB symptoms undergoing intradetrusor injection of 200 units (or more) of BTX-A will be more willing to pursue additional sessions of BTX-A injections with a protocol utilizing less injection sites, while still maintaining effectiveness of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women (>18 years of age) with a diagnosis of neurological conditions such as MS, PD, CVA, myelomeningocele, SCI, or traumatic brain injury longer than 6 months prior to treatment.
* Diagnosis of neurogenic bladder indicated for treatment with BTX-A for OAB symptoms.
* Participants must be able to provide informed consent, as well as understand and be willing to undergo.

follow-up procedures and completion of all questionnaires provided during the study.

Exclusion Criteria:

* Symptomatic UTI at the time of procedure, defined as positive nitrites or high-volume leukocyte esterase on urine dip in addition to at least one of the following symptoms: dysuria, gross hematuria, suprapubic pain, frequency/urgency above baseline.
* Diagnosis of bladder pain syndrome or other chronic pain syndrome including fibromyalgia, chronic pelvic pain, pelvic floor dysfunction, levator myalgia.
* Untreated bladder malignancy.
* Women who are currently pregnant or breast feeding.
* Contraindications to intradetrusor BTX-A injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rose Khavari, MD, Principal Investigator — Houston Methodist Research Group
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen A, Stewart J, Gonzalez RR, Stampas A, Kobashi K, Khavari R. Optimizing the Injection Schema for Higher Doses of OnabotulinumtoxinA (BTX-A) in the Office Setting: A Randomized Prospective Trial for Patients With Neurogenic Lower Urinary Tract Dysfunction and Idiopathic Overactive Bladder. Neurourol Urodyn. 2025 Nov;44(8):1537-1544. doi: 10.1002/nau.70130. Epub 2025 Aug 20. PMID 40836399

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Injection Sites | Reduced Injection Sites
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Initially, 78 patients met the inclusion criteria and provided consent. Two were later excluded: one due to urinary tract infection symptoms and a suspicious urinalysis, and the other due to severe autonomic dysreflexia, which was identified after consent but before the procedure. The physician deemed the procedure unsafe in the clinic setting, leading to exclusion.
Groups:
- Standard Injection Sites (20): Standard number of injection sites: 200 units or 300 units BTX-A reconstituted in 20 mL normal saline, injected into the bladder detrusor in 20 separate injections of 1 mL including the trigone.
- Reduced Injection Sites (5): Reduced number of injection sites: 200 units or 300 units BTX-A reconstituted in 5 mL normal saline, injected into the bladder detrusor in 5 separate injections of 1 mL including the trigone.
- Total: Total of all reporting groups
Arm/Group | Standard Injection Sites (20) | Reduced Injection Sites (5) | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (22.2) | 47.7 (19.4) | 48.95 (20.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 8 | 11 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 27 | 33 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Medical comorbidities [Number; unit: participants]
  Multiple Sclerosis | 8 | 7 | 15
  Sacral Agenesis | 1 | 1 | 2
  Spina Bifida | 15 | 11 | 26
  Spinal Cord Injury | 4 | 11 | 15
  Cerebral Vascular Accident | 1 | 4 | 5
  Parkinsons Disease | 1 | 0 | 1
  Chronic Inflammatory Demyelinating Polyneuropathy | 1 | 0 | 1
  Syringomyelia | 0 | 1 | 1
  Transverse Myelitis | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Willingness to Repeat Procedure
Description: Participants were asked to rate their willingness to repeat the procedure using an 11-point visual analog scale (VAS). A score of 0 ("Never") indicates complete unwillingness, representing the least favorable outcome, while a score of 11 ("Definitely") reflects strong willingness, representing the most favorable outcome.
Time Frame: Immediately post-procedure and 6 weeks post-procedure
Population: Data at 6-weeks post-procedure were available for 54 participants. Loss to follow-up included 10 participants from the 20-injection group and 12 participants from the 5-injection group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard Injection Sites (20): 200 units or 300 units BTX-A reconstituted in 20 mL normal saline, injected into the bladder detrusor in 20 separate injections of 1 mL including the trigone.
- Reduced Injection Sites (5): 200 units or 300 units BTX-A reconstituted in 5 mL normal saline, injected into the bladder detrusor in 5 separate injections of 1 mL including the trigone.
Arm/Group | Standard Injection Sites (20) | Reduced Injection Sites (5)
Number analyzed (Participants) | 38 | 38
units on a scale
  Post-injection willingness to repeat procedure rating (VAS score) | 9.16 (1.46) | 9.34 (1.26)
  6-weeks post-procedure willingness to repeat procedure rating (VAS score): number analyzed (Participants) | 28 | 26
  6-weeks post-procedure willingness to repeat procedure rating (VAS score) | 9.73 (1.12) | 9.67 (0.99)
Statistical Analysis 1: Comparison: Standard Injection Sites (20) vs Reduced Injection Sites (5); Willingness to repeat procedure immediately after received intradetrusor BTX-A injections; Test type: Other; p = 0.57, t-test, 2 sided — Threshold for statistical significance used P-value <0.05
Statistical Analysis 2: Comparison: Standard Injection Sites (20) vs Reduced Injection Sites (5); Willingness to repeat procedure asses 6-weeks after intradetrusor BTX-A injections; Test type: Other; p = 0.83, t-test, 2 sided — Threshold for statistical significance used P-value <0.05

2. Secondary Outcome: Change in Neurogenic Bladder Symptoms After BTX-A Treatment - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF)
Description: The ICIQ-SF is a standardized survey that assesses the frequency, severity, and impact of urinary incontinence (UI) on quality of life (QoL). The total score, ranging from 0 to 21, is calculated from three questions, with higher scores indicating more severe symptoms. A score of 0 reflects no leakage and no impact on QoL. Question 1 measures how often leakage occurs (0-5), Question 2 assesses the amount of leakage (0-6), and Question 3 evaluates the impact on QoL (0-10), with higher scores indicating worse outcomes. We report the mean difference in total ICIQ and QoL scores from baseline to 6-weeks post-treatment.
Time Frame: Baseline and 6-weeks after BTX-A injections
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Injection Sites (20) | Reduced Injection Sites (5)
Number analyzed (Participants) | 28 | 26
units on a scale
  Mean difference in Total ICIQ score | -4.11 (8.25) | -5.23 (6.55)
  Mean difference in ICIQ QoL score | -2.33 (4.38) | -3.54 (3.70)
Statistical Analysis 1: Comparison: Standard Injection Sites (20) vs Reduced Injection Sites (5); Difference in total ICIQ-SF score assessed before and 6-weeks after treatment; Test type: Other; p = 0.59, t-test, 2 sided — Threshold for statistical significance used P-value <0.05
Statistical Analysis 2: Comparison: Standard Injection Sites (20) vs Reduced Injection Sites (5); Difference in ICIQ QoL score assessed before and 6-weeks after treatment; Test type: Other; p = 0.29, t-test, 2 sided — Threshold for statistical significance used P-value <0.05

3. Secondary Outcome: Change in Neurogenic Bladder Symptoms After BTX-A Treatment - Neurogenic Bladder Symptom Score - Short Form (NBSS-SF)
Description: The NBSS-SF is a validated survey with 10 questions that measure bladder symptoms across 3 different domains: incontinence (score range: 0-12), storage and voiding (score range: 0-9), and consequences (score range: 0-7); the highest score is associated with worse symptoms. It also includes one question to assess overall quality of life (QoL) scored from 0 (pleased) to 4 (unhappy). The total score, ranging from 0 to 28, is calculated from the three domains (Q3-Q10), with 0 being the best outcome and 28 the worst outcome. Here we report the mean difference in total NBSS-SF, each of the domains and QoL scores from baseline to 6-weeks post-treatment.
  The NBSS-SF is a validated 10-question survey that assesses bladder symptoms across three domains: incontinence (score range: 0-12), storage and voiding (score range: 0-9), and consequences (score range: 0-7), with higher scores indicating worse symptoms. It also includes a quality of life (QoL) question (Q2) scored from 0 (pleased)
Time Frame: Baseline and 6-weeks after BTX-A injections
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Injection Sites (20) | Reduced Injection Sites (5)
Number analyzed (Participants) | 28 | 26
units on a scale
  Mean difference in Total NBSS-SF | 5.44 (4.19) | 4.65 (5.46)
  Mean difference in NBSS-SF QoL | -1.81 (1.54) | -2.15 (1.46)
  Mean difference in NBSS-SF incontinence domain | -2.93 (2.92) | -2.15 (1.46)
  Mean difference in NBSS-SF storage and voiding domain | -2.96 (2.47) | -3.04 (3.39)
  Mean difference in NBSS-SF consequence domain | -2.63 (2.41) | -3.00 (3.19)
Statistical Analysis 1: Comparison: Standard Injection Sites (20) vs Reduced Injection Sites (5); Difference in total NBSS-SF score assessed before and 6-weeks after treatment; Test type: Other; p = 0.57, t-test, 2 sided — Threshold for statistical significance used P-value <0.05
Statistical Analysis 2: Comparison: Standard Injection Sites (20) vs Reduced Injection Sites (5); Difference in NBSS-SF QoL score assessed before and 6-weeks after treatment; Test type: Other; p = 0.42, t-test, 2 sided — Threshold for statistical significance used P-value <0.05
Statistical Analysis 3: Comparison: Standard Injection Sites (20) vs Reduced Injection Sites (5); Difference in NBSS-SF incontinence domain score assessed before and 6-weeks after treatment; Test type: Other; p = 0.24, t-test, 2 sided — Threshold for statistical significance used P-value <0.05
Statistical Analysis 4: Comparison: Standard Injection Sites (20) vs Reduced Injection Sites (5); Difference in NBSS-SF storage and voiding domain score assessed before and 6-weeks after treatment; Test type: Other; p = 0.93, t-test, 2 sided — Threshold for statistical significance used P-value <0.05
Statistical Analysis 5: Comparison: Standard Injection Sites (20) vs Reduced Injection Sites (5); Difference in NBSS-SF consequences domain score assessed before and 6-weeks after treatment; Test type: Other; p = 0.64, t-test, 2 sided — Threshold for statistical significance used P-value <0.05

4. Secondary Outcome: Patient Impression of Clinical Improvement After BTX-A - Patient Global Impression of Improvement (PGI-I) Scale
Description: The PGI-I is a validated tool for assessing patient satisfaction after therapy. It consists of a single question using a Likert scale to measure perceived improvement or worsening after BTX-A treatment, ranging from 1 ("Very much worse") to 7 ("Very much better"). Data reported here reflect average scores obtained at the six-week follow-up.
Time Frame: 6 weeks after BTX-A injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Injection Sites (20) | Reduced Injection Sites (5)
Number analyzed (Participants) | 28 | 26
units on a scale | 5.26 (1.04) | 4.88 (1.09)
Statistical Analysis 1: Comparison: Standard Injection Sites (20) vs Reduced Injection Sites (5); Test type: Other; p = 0.21, t-test, 2 sided — Threshold for statistical significance used P-value <0.05

5. Secondary Outcome: Patient Reported Procedural Discomfort - Numeric Pain Rating Scale (NPRS)
Description: Participants rated their pain using the NPRS to assess discomfort during the BTX-A procedure. The NPRS is an 11-point scale (0-10), where 0 represents no pain and 10 indicates the worst pain ever experienced. Higher scores reflect greater pain intensity. We report the change in NPRS scores from before to immediately after the procedure.
Time Frame: Prior to and immediately after BTX-A injections
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Injection Sites (20) | Reduced Injection Sites (5)
Number analyzed (Participants) | 38 | 38
units on a scale | 3.39 (3.01) | 0.57 (2.07)
Statistical Analysis 1: Comparison: Standard Injection Sites (20) vs Reduced Injection Sites (5); Change in post-procedural pain as compared to baseline; Test type: Other; p < 0.00002, t-test, 2 sided — Threshold for statistical significance used P-value <0.05

ADVERSE EVENTS:
Time Frame: 6-8 weeks post-injection
Groups:
- Standard Injection Sites (20): Standard number of injections (20 injections): 200 units or 300 units BTX-A reconstituted in 20 mL normal saline, injected into the bladder detrusor in 20 separate injections of 1 mL including the trigone.
- Reduced Injection Sites (5): Reduced number of injections (5 injections): 200 units or 300 units BTX-A reconstituted in 5 mL normal saline, injected into the bladder detrusor in 5 separate injections of 1 mL including the trigone.
Arm/Group | Standard Injection Sites (20) | Reduced Injection Sites (5)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 7/28 | 8/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Injection Sites (20) (N=28) | Reduced Injection Sites (5) (N=26)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 6 (6) | 7 (7)
Catheter Clogging (Renal and urinary disorders) | 0 (0) | 1 (1)
New onset gross hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Increased bladder spasms (Renal and urinary disorders) | 0 (0) | 1 (1)
Decreased cold tolerance (Endocrine disorders) | 0 (0) | 1 (1)
Hyperglycemia requiring emergency evaluation (Endocrine disorders) | 1 (1) | 0 (0)
Plasmapheresis for CIDP (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT06059066/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT06059066/ICF_001.pdf